CLINICAL TRIAL: NCT02288923
Title: A Randomised, Observer Blinded, Controlled Trial Of Femoral Nerve Block Versus Local Infiltration Analgesia for Post Operative Analgesia Following Total Knee Arthroplasty
Brief Title: Trial to Compare Femoral Nerve Block With Local Anaesthetic Injection for Post-operative Pain After Knee Replacement.
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Fiona Martin, Consultant Anaesthetist, Royal Devon and Exeter NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14/SW/0016; 139814 (Other: IRAS Number)
Record Dates: First submitted 2014-11-04; First posted 2014-11-13 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Arthritis Knee
Keywords: Total knee arthroplasty; Femoral nerve block; Local infiltration analgesia
MeSH Terms: interventions — Anesthesia, General; Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral nerve block (Active Comparator): Femoral nerve block with 20ml 0.375% Levobupivacaine
  Interventions: Procedure: Femoral nerve block; Procedure: Sub arachnoid analgesia; Procedure: Sedation or general anaesthesia; Drug: Pre-medication; Drug: Intra-operative medication; Drug: Post-operative analgesia - morphine; Drug: Post-operative analgesia - ibuprofen and paracetamol; Drug: Regular anti emetics
- Local Infiltration Analgesia (Active Comparator): Local infiltration of knee joint using 40ml of bupivacaine 0.25% with adrenaline 1:200 000, diluted to 150ml with saline 0.9%. This is then divided into thirds; 50ml into the posterior capsule before cementing, 50ml into the medial and lateral capsules and 50ml into subcutaneous tissues and in and around the vastus medialis and sartorius muscles (where it may block the saphenous nerve).
  Interventions: Procedure: Local Infiltration Analgesia; Procedure: Sub arachnoid analgesia; Procedure: Sedation or general anaesthesia; Drug: Pre-medication; Drug: Intra-operative medication; Drug: Post-operative analgesia - morphine; Drug: Post-operative analgesia - ibuprofen and paracetamol; Drug: Regular anti emetics

INTERVENTIONS:
Procedure: Femoral nerve block — Supine position
  If using peripheral nerve stimulator for localisation of the femoral nerve:
  50 mm insulated needle Peripheral nerve stimulator set at 2 Hz with pulse width 100μs When quadriceps muscle twitch is present with a stimulated current between 0.2 and 0.5mA, inject 20ml 0.375% (3.75mg/ml) Levo- bupivacaine
  If using ultrasound for localisation of the femoral nerve:
  High frequency linear array probe Short bevelled nerve-block needle, using in or out of plane technique Inject 20ml 0.375% (3.75mg/ml) Levo-bupivacaine underneath fascia iliaca ensuring adequate spread of local anaesthetic
  Other Names: Femoral nerve blockade; Regional anaesthesia femoral nerve
  Arms: Femoral nerve block
Procedure: Local Infiltration Analgesia — Local infiltration analgesia to be administered by surgeon towards the end of operation:
  40ml of bupivacaine 0.25% with adrenaline 1:200 000, diluted to 150ml with saline 0.9%. This is then divided into thirds; 50ml into the posterior capsule before cementing, 50ml into the medial and lateral capsules and 50ml into subcutaneous tissues and in and around the vastus medialis and sartorius muscles (where it may block the saphenous nerve).
  Other Names: LIA
  Arms: Local Infiltration Analgesia
Procedure: Sub arachnoid analgesia — Patients in both arms of the trial will be given sub arachnoid anasthesia of 2.5-3.0ml of plain bupivacaine 0.5% using a 25G Whitacre needle. Patients may have 0-4mg midazolam and/or 0-1mcg/kg fentanyl and/or 0-4mcg/ml propofol sedation using the Marsh protocol if required for this procedure as deemed appropriate by the anaesthetist.
Procedure: Sedation or general anaesthesia — After insertion of the sub arachnoid anaesthesia the patient may choose to be fully asleep or sedated. If they choose to be fully asleep, they may have up to 2mcg/kg fentanyl in total (including any given at time of subarachnoid injection), muscle relaxation as indicated for facilitation of intubation where needed, airway control using LMA or tracheal tube where needed, and general anaesthesia maintained using inspired oxygen concentration of 0.3-0.7 with propofol up to 5mcg/kg (Marsh protocol) or isoflurane or sevoflurane. If the patient chooses to have sedation they may have additional midazolam up to a total dose of 4mg and/or a propofol infusion (Marsh protocol) of 0-4mcg/ml.
Drug: Pre-medication — All patients will receive 1g paracetamol pre-operatively. Those on non steroidal anti inflammatory drugs may continue to take them. Apart from these, no other pain relieving pre-medications are to be used. Patients may be given anxiolysis using temazepam 10-20mg or diazepam 2-5mg by mouth if required. Antacid premedication is permitted using ranitidine, metoclopramide or proton pump inhibitors.
Drug: Intra-operative medication — If paracetamol has not been given pre-operatively, it will be given intraoperatively 1g IV. Where 2 or more of the following risk factors are present; female, non smoker, previous post operative nausea or vomiting, intra operative opiates, the patients will be given 4mg dexamethasone and or 4mg ondansetron IV. Vasopressor drugs may be given at the anaesthetist's discretion to maintain an appropriate blood pressure. Intraoperative fluid infusion is at the discretion of the anaesthetist. Antibiotic prophylaxis is as per the hospital protocol (currently 6mg/kg Teicoplanin IV and 3mg/kg gentamicin pre induction). Tranexamic acid will be given as per unit protocol, (currently 1g pre-operatively IV and 500mg orally at 8 hours post op. unless contraindicated by a high risk of thrombosis.)
Drug: Post-operative analgesia - morphine — Patients will all be given a morphine pump which will give 1mg every 5 minutes. This is to be discontinued after 48 hours and changed to oral morphine 10-20mg if weight 50-70kg, 20-30mg if weight >70kg 2 hourly.
Drug: Post-operative analgesia - ibuprofen and paracetamol — All patients will be given 1g paracetamol 6 hourly and 400mg ibuprofen 8 hourly unless there are contraindications. If patients are on an alternative non-steroidal anti inflammatory drug then this may be substituted for ibuprofen.
Drug: Regular anti emetics — All patients will receive 4mg ondansetron regularly for 2 days. They will be prescribed 50mg cyclizine as an addition to this if needed.

SUMMARY:
Pain after a knee replacement can impair recovery and use of the new knee. Having an injection to numb the femoral nerve is known to give good pain relief after the operation but may lead to slower mobilisation as it also prevents the patient from moving the knee. Recent studies have shown that infiltration of local anaesthetic (LIA) within the new knee joint may also give good pain relief. The null hypothesis is that there is no difference in primary or secondary outcome measures between femoral nerve block and LIA, as anaesthetic techniques for knee replacement.

DETAILED DESCRIPTION:
Knee pain and stiffness is a common problem which can sometimes be improved by inserting a replacement knee joint. An anaesthetist is a doctor who specialises in looking after patients undergoing surgery, and there are a variety of different anaesthetics which can be used for knee replacement surgery. These include general anaesthesia (going to sleep), and spinal or epidural anaesthesia (where pain killers are injected into the back, resulting in temporarily numb legs). Pain killers can also be injected around the nerves which supply the leg, or around the site of the operation itself, combined with general or spinal anaesthesia if required.

Over the years, multiple different combinations of these techniques have been tried. All have advantages and disadvantages. Generally, those which completely numb the leg after the operation often cause weakness which interferes with movement. Although the patient will have no pain, getting up and around with the physiotherapist is crucial and the weakness can delay recovery. However, excessive pain can also interfere with movement. There is therefore a balance to be struck between pain and weakness, and the choice of anaesthetic technique is key.

Researchers previously conducted a study at the Royal Devon and Exeter Hospital which compared the effects of two techniques; the use of diamorphine in a spinal injection, and the injection of pain killer around a nerve supplying the leg (femoral nerve block, FNB). Whilst the research showed that FNB gave better pain relief, there are still concerns that it causes weakness which may interfere with movement. A newer technique has evolved over recent years in which pain killer is injected directly around the knee during the operation. This is known as local infiltration analgesia (LIA) and the potential advantages are that it is simple, safe and does not cause leg weakness.

If research shows that LIA provides adequate pain relief without weakness, it may be a better option to use routinely, rather than FNB. The primary outcome measure is the amount of morphine used in the first 48 hours. The secondary outcome measures are the Total Pain Relief Score (TOTPAR), post operative pain scores, the ability to achieve set rehabilitation goals, readiness for discharge and qualitative data on patient recovery and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

All adult patients presenting for primary knee arthroplasty under the care of the Exeter Knee Unit Consultants Messrs Toms, Eyres, Cox, Mandalia, Schrantz.

Exclusion Criteria:

1. Total knee arthroplasty for trauma
2. Unicompartmental surgery
3. Bilateral surgery
4. Contra indication to spinal anaesthesia or peripheral nerve blocks (anticoagulation, hydrocephalus, raised intracranial pressure, peripheral neuropathy)
5. Allergy to local anaesthetics or morphine
6. Chronic pain:

   * Under active follow up by chronic pain team
   * Chronic strong opiate use (morphine, oxycodone, buprenorphine, pethidine, methadone). Codeine, dihydrocodeine and tramadol are not included
   * Other chronic pain medications (including gabapentin, pregabalin or amitriptyline)
7. Unable to adequately understand verbal explanations or written information given in English, or patients with special communication needs -

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in first post-operative 72 hours | 72 hours
  The total amount of morphine consumed by the patient in the first 72 post-operative hours will be added up. If morphine has been given orally it will be counted as ⅓ the intravenous dose.

SECONDARY OUTCOMES:
Total pain relief score | Post op days 1, 2 and 3
  Using the TOTPAR Scoring system (40. Cooper SA, and Beaver WT. A model to evaluate mild analgesics in oral surgery outpatients. Clin Pharmacol Ther. 1976, Aug;20(2):241-50.), patients will have their overall time measured when their pain was 70% controlled during post operative days 1, 2 and 3.
Post operative pain scores | Day 0 - 3 post op
  Pain scores (using the numerical rating scale of 0-10) will be collected from patients at 12, 24, 48 and 72 hours post operation. A significant reduction would be a decrease of pain score at any of these times of 1.5 or more.
Achievement of rehabilitation goals | 1-4 days post operatively
  Ability to achieve the rehabilitation goals of standing and getting out into a chair on post op day 1, walking to the bathroom at the end of day 2 and walking independently with crutches by the end of day 4
Readiness for discharge | Post operative day 2-10
  Time when patient is ready for discharge from the acute care hospital.
Patient satisfaction | 2nd post-operative day
  Patients will be asked to fill out a patient satisfaction questionnaire "quality of recovery 40" (QoR-40) Myles PS, Weitkamp B, Jones K, Melick J, and Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. British Journal of Anaesthesia. 2000;84(1):11-15.
Oxford Knee Score | Pre op and 6 weeks post operatively
  The Oxford Knee score will be completed by patients before and 6 weeks after their operation. http://www.orthopaedicscore.com/scorepages/oxford_knee_score.html
EuroQol 5 dimensions score | Pre op and 6 weeks post operatively
  EQ-5D-5L (EuroQol 5 dimensions score) will be used to measure the satisfaction the patient has with their knee in the fields of mobility, self-care, usual activities, pain/discomfort and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Martin, MBCHB, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon, United Kingdom